CLINICAL TRIAL: NCT07206030
Title: FRiEND Registry: Real Life Data From Hypertensive Patients Treated With Renal Denervation in Current Practice in France- French RENal Denervation Registry
Brief Title: Real Life Data From Hypertensive Patients Treated With Renal Denervation in Current Practice in France- French RENal Denervation Registry
Acronym: FRIEND
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC25.0159; 23540206 (Other: Health Data Hub)
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Hypertension (HTN)
Keywords: Hypertension (HTN); RDN; Renal denervation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Renal denervation (RDN) is a recent procedure that can be used to control BP (blood pressure) in hypertensive patients. Numerous publications from randomised trials have demonstrated the efficacy of RDN in this indication. The latest guidelines now include RDN as an effective technique for use in hypertension. Since early 2023, RDN using Medtronic's Spiral radiofrequency system has benefited from transitional authorisation for reimbursement by the French health insurance system. An application for reimbursement is underway for the ultrasound system. We aim to compile an exhaustive prospective register of all procedures carried out in France over the next few years, regardless of the type of catheter used or the context in which the procedure was carried out (transitional reimbursement, industrial register, randomised trial). Our aim is to assess the efficacy and safety of the procedure within the French healthcare system, the characteristics of patients benefiting from the procedure, the centres performing renal denervation, and the care pathways used, and to be able to present all this data, independently of the industry, to the healthcare authorities when it comes time to reassess the value of this procedure and its indications. The goal of this observational study is to learn about changes in blood pressure in patient with high blood pressure before and 1 year after a renal denervation treatment (RDN).

The primary endpoint is to describe changes in systolic blood pressure (SBP) measured by Home Blood Pressure Measurement (HBPM) in patients suffering from high blood pressure, before and 1 year after RDN.

DETAILED DESCRIPTION:
This study concerns patients with high blood pressure who have been treated with renal denervation since January 2010 or who will undergo renal denervation after March 2025.

ELIGIBILITY:
Inclusion Criteria:

* Adult ( > 18 years old) hypertensive patients treated with RDN in France whatever the catheter and the indication. This might include retrospective data for patient already treated with RDN in the past.

Exclusion Criteria:

* RDN not proposed to the patient, patient opposing the collection and use of his/her data for research purposes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a confirmed diagnosis of high blood pressure, eligible for a renal denervation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in SBP measured by HBPM before and after RDN (1 year). | before intervention and 1 year after intervention
  Measurement of home blood pressure before and 1 year after RDN

SECONDARY OUTCOMES:
Evaluate changes in office systolic blood pressure using the combination of SBP measured in HBPM and 24-hour-Automatic Blood Pressures Measurements (ABPM) before, 3 months, 6 months and 1 year, after DNR treatment. | before the DNR intervention and 3, 6, 12 months after DNR intervention
  collection of home systolic blood pressures and 24-hour-Automatic Blood Pressures Measurements before, 3 months, 6 months and 1 year, after DNR treatment.
Evaluate the evolution at 3 months, 6 months, 1 year, of the drug burden in antihypertensive treatment, the percentage of patients having reached the blood pressure target and the win ratio. | Before intervention and 1-3, 6, 12 months after DNR intervention
  Collection of treatments taken by the patient and des Blood pressures values
Evaluate the development of renal artery stenosis before and 6 months, 1 year, after DNR. | before DNR, 6, 12 months after DNR
  Appearance of renal artery stenosis on Renal Arteries ultrasound or Renal arteries CT angiography images
Evolution of creatinine levels before and 6 months, 1 year, after DNR. | before, 6 and 12 months after DNR
  collection of blood creatinine value
Evaluate the occurrence of other complications related to hypertension or to the procedure itself | from DNR intervention to 1 year follow up
  Collection of adverse events and complications after DNR
Comparison of responders and non-responders to the procedure (24h ABPM systolic blood pressure decrease of 5 mmHg or more and/or the diminution of the medical burden by at least one therapeutic class without SBP increase compared to baseline). | inclusion, 1, 6, 12 months after the DNR procedure
  Collection of systolic blood pressure measurements and medical treatment from inclusion to 1 year after the DNR procedure.
Evaluate the performance of known predictors of response to renal denervation in our population. | from inclusion to 1 year follow up after the procedure
  To investigate how well known predictors of response to renal denervation work in patients in our group
Describe the type of center performing the procedure, the context in which DNR is performed, patient characteristics and care pathways. | from inclusion to 1 year follow-up
  Collection of type of center performing the DNR procedure, the indication for the DNR procedure, patient characteristics and care pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier ORMEZZANO, Doctor of medicine, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Chu Grenoble Alpes, La Tronche, France, France

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2025-04-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT07206030/Prot_000.pdf